CLINICAL TRIAL: NCT03801720
Title: UltraWee: Ultrasound Bladder Stimulation to Help With Clean Catch Urine in Pre-Continent Children
Brief Title: UltraWee: Ultrasound Bladder Stimulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was suspended due to COVID. Investigators no long feel that completion of the study is feasible and have permanently terminated the study.
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Vincent Calleo, Principal Investigator, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1190457
Record Dates: First submitted 2018-12-14; First posted 2019-01-11 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Urinalysis
Keywords: Clean Catch Urine (CCU); Catherterization; Ultrasound; Micturition; Urine Collection; Pre-Continent Children; Pediatrics
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Utilize standard practice for obtaining a CCU in pre-continent children; this consists of cleaning the GU area with betadine and waiting 5 minutes for micturition to occur.
- Experimental Group (Experimental): Consists of cleaning the GU area with betadine followed by using an ultrasound probe to apply cool ultrasound gel and subprapubic pressure to the patient to induce micturition.
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Using ultrasound stimulation to induce micturition.
  Arms: Experimental Group

SUMMARY:
The UltraWee study is a prospective randomized controlled trial used to compare the success rate of and time to obtaining a urine sample in pre-continent children between standard clean catch urine (CCU) method and using ultrasound stimulation clean catch methods. The objectives of this study are to see if ultrasound stimulation increases success rate of micturition, decreases time to micturition, and decreases the use of more invasive techniques for urine collection.

DETAILED DESCRIPTION:
Standard procedure for obtaining urine samples in the pediatrics emergency department consists of a clean catch urine (CCU). For those patients who are still pre-continent, this involves cleaning the genitourinary (GU) area with betadine followed with waiting with a specimen cup for the patient to produce urine.

Currently, the CCU technique has had mixed success rates of micturition, some studies showing as low as 12% success rate. Because of the mixed success rates, often times these patients are subjected to the discomfort and trauma of a urinary catheter. Catheterization also occurs in patients with clinical conditions that require urine samples under time sensitive conditions.

Less invasive ways of urine collections have been recently studied. The Quick-Wee study was a novel study that showed a promising alternative to obtaining urine samples in pre-continent children when compared to the CCU sample. This method served as a noninvasive way to obtain a urine sample, thus preventing uncomfortable and traumatic urinary catheterizations and improving parent satisfaction scores.

The investigators hope to study the effectiveness of another technique for obtaining a urine sample without urinary catheterization: ultrasound stimulation. By incorporating ultrasound evaluation of the bladder, the UltraWee study hopes to decrease the number of failed attempts at obtaining a urine sample in pre-continent children less than thirty-six months of age.

The UltraWee study will be a prospective randomized controlled trial comparing success rate of and time to obtaining a urine sample in pre-continent children between standard clean catch urine method and using ultrasound stimulation clean catch methods. The objective of this study is to see if ultrasound stimulation increases success rate and decreases time to micturition.

ELIGIBILITY:
Inclusion Criteria:

* Pre-continent children
* Children between the ages of 1 month and 36 months
* Children who require a urine sample as part of their workup
* Children who are seen in the emergency department at University Hospital Downtown Campus

Exclusion Criteria:

* Children who are continent
* Children who are in foster care or who are wards of the state

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Incidence of miturition | Less than 5 minutes
  Recorded act of successfully initiating miturition/urination
Time to Miturition | 0-5 minutes
  Recorded time to miturition

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Calleo, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No